CLINICAL TRIAL: NCT00355875
Title: Oxygen Exposure During Newborn Resuscitation and Pulmonary Oxidative Stress
Brief Title: The Effect of Oxygen Exposure During Newborn Resuscitation on Lung Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Equipment loan from Masimo Corp. (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RT754957
Record Dates: First submitted 2006-07-22; First posted 2006-07-25 (Estimated); Last update posted 2006-11-07 (Estimated); Status verified 2006-11

CONDITIONS: Prematurity; Oxidative Pulmonary Injury
Keywords: newborn; preterm; resuscitation; oxidative injury; protein carbonyl
MeSH Terms: conditions — Premature Birth

INTERVENTIONS:
Procedure: titration of oxygen during resuscitation

SUMMARY:
Hypothesis: In this feasibility study, hyperoxemia, as approximated by transcutaneous hemoglobin saturation with oxygen (Sp02), at the time of birth will cause sustained pulmonary oxidative stress as demonstrated by elevation of pulmonary protein carbonyl. Furthermore, this oxidative stress will be directly proportional to the imposed oxygen-burden during resuscitation at the time of birth.

This study will give us information regarding the magnitude of protein carbonyl elevation in the preterm infant. With these results we will be able to 1. establish the technique for the running or protein carbonyl assays and 2. calculate an appropriate sample size for a future randomized control trial.

DETAILED DESCRIPTION:
Immediately prior to birth, preterm infants (<= 32 weeks gestation) will be randomized to one of three groups: 1. Low Oxygen Burden (LOB) - initiation of resuscitation with 21% 02, II. Moderate Oxygen Burden (MOB) - initiation of resuscitation with 100% 02 and III. High Oxygen Burden (HOB) - 100% 02 used for the entire resuscitation. A pulse oximetry monitor will be connected to a probe on the infant's hand to measure the transcutaneous hemoglobin saturation with oxygen (Sp02). Adjustments to the inspired oxygen concentration will be made every 15 seconds for infants in the LOB and MOB groups to achieve a target Sp02 range of 85-92%. Resuscitation will otherwise proceed as per standard of care. The intervention will end upon arrival in the neonatal intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* <=32 weeks gestation
* inborn
* require intubation

Exclusion Criteria:

* lethal anomalies
* cyanotic congenital heart disease
* known hemoglobinopathy
* risk factors for persistent pulmonary hypertension

Ages: 23 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30
Dates: Start 2005-07; Study Completion 2006-10

PRIMARY OUTCOMES:
protein carbonyl concentration in the tracheal aspirate on day 1

SECONDARY OUTCOMES:
protein carbonyl concentration in the tracheal aspirate on day 3
protein carbonyl concentration in the tracheal aspirate on day 7
protein carbonyl concentration in the tracheal aspirate on day 14
protein carbonyl concentration in the tracheal aspirate on day 21
protein carbonyl concentration in the tracheal aspirate on day 28

CONTACTS AND LOCATIONS:
Overall Officials: Yacov Rabi, MD, FRCPC, Principal Investigator — University of Calgary
Locations (1):
- Canada, Calgary, Alberta, Canada